CLINICAL TRIAL: NCT01953783
Title: A Phase 1 Study of [ 14 C]-Ixazomib to Assess Mass Balance, Pharmacokinetics, and Metabolism in Patients With Advanced Solid Tumors or Lymphoma
Brief Title: Mass Balance, Pharmacokinetics and Metabolism Study of IXAZOMIB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C16016
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Results first posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Advanced Solid Tumors; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IXAZOMIB (Experimental): Part A: Participants will receive a single dose of 4.1-milligram (mg) [14C]-IXAZOMIB oral solution containing approximately 500-nCurie (nCi) of total radioactivity on Day 1 and remain at the clinic for 8 days. On Days 14 and 21, participants may be administered a single 4.0-mg capsule of IXAZOMIB. Participants will return to the clinic in the evening before Days 14, 21, 28, and 35 for a 24-hour overnight clinic visit.
  Part B: Eligible participants from Part A may continue into Part B once they have completed their Day 35 assessments in Part A. Participants may receive IXAZOMIB capsules administered orally at a dose of 4.0-mg once weekly on Days 1, 8, and 15 of 28-day cycles. Participants will continue in this study until disease progression or unacceptable toxicity.
  Interventions: Drug: IXAZOMIB

INTERVENTIONS:
Drug: IXAZOMIB — Part A: Ixazomib 4.1 mg containing approximately 500-nCi [14C]-ixazomib, solution, orally on Day 1 and ixazomib 4 mg, capsule, orally on Days 14 and 21.
  Part B: Ixazomib 4 mg, capsule, orally, once weekly, on Days 1, 8 and 15 in 28-day cycles until disease progression or unacceptable toxicity.

SUMMARY:
This is a phase 1, 2-part, open-label study in 4 to 6 pharmacokinetic-evaluable participants with advanced solid tumors or lymphoma.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all of the following inclusion criteria to be enrolled in the study:

* 18 years or older
* Histologic or cytologic diagnosis of advanced or metastatic solid tumor or lymphoma for which no standard, curative, or life-prolonging therapies exist or are effective
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Female participants who are postmenopausal for at least 1 year OR are surgically sterile OR if of childbearing potential, agree to practice 2 effective methods of contraception at the same time during the entire study through 90 days after the last dose of study drug OR agree to practice true abstinence
* Male participants who agree to practice effective barrier contraception during the entire study and through 90 days after the last dose of study drug OR agree to practice true abstinence
* Voluntary written consent
* Suitable venous access for the conduct of blood sampling
* Recovered from the reversible effects of prior anticancer therapy

Exclusion Criteria:

Participants meeting any of the following exclusion criteria are not to be enrolled in the study:

* Female participants who are lactating or breastfeeding or have a positive serum pregnancy test
* Serious medical or psychiatric illness that could interfere with the study
* Treatment with any investigational products or radiotherapy within 21 days before the first dose of study drug
* Peripheral neuropathy greater than (>) Grade 2
* Systemic treatment with strong and moderate inhibitors of CYP1A2, strong and moderate inhibitors of CYP3A, or clinically significant CYP3A inducers or use of Ginkgo biloba or St. John's wort within 14 days before the first dose of study drug
* Symptomatic brain metastasis. Participants with brain metastases: must have stable neurologic status following local therapy (surgery or radiation) for at least 2 weeks after completion of the definitive therapy; and must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events (AEs)
* Ongoing treatment with corticosteroids
* Major surgery within the 14 days preceding the first dose of study drug
* Infection requiring systemic intravenous antibiotic therapy or other serious infection within 14 days before the first dose of study drug
* Life-threatening illness unrelated to cancer
* Known hepatitis B surface antigen -positive, or known or suspected active hepatitis C infection or human immunodeficiency virus (HIV) positive
* Diagnosed or treated for another malignancy within 2 years before the first dose, OR previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
* Any cardiovascular condition specified in the study protocol
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of IXAZOMIB
* History of urinary and/or fecal incontinence
* Inability to comply with study procedures or visit schedule including the requirement for inpatient confinement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-03-19 (Actual); Primary Completion 2014-12-17 (Actual); Study Completion 2016-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Cleveland, Ohio, United States

REFERENCES:
- [Derived] Gupta N, Zhang S, Pusalkar S, Plesescu M, Chowdhury S, Hanley MJ, Wang B, Xia C, Zhang X, Venkatakrishnan K, Shepard DR. A phase I study to assess the mass balance, excretion, and pharmacokinetics of [14C]-ixazomib, an oral proteasome inhibitor, in patients with advanced solid tumors. Invest New Drugs. 2018 Jun;36(3):407-415. doi: 10.1007/s10637-017-0509-1. Epub 2017 Sep 21. PMID 28932928

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 19 March 2014 to 09 February 2016.
Pre-assignment Details: Participants with a historical diagnosis of advanced solid tumors or lymphoma were enrolled in 1 treatment group of this 2-part study to receive ixazomib.
Groups:
- Ixazomib: Ixazomib 4.1 milligram (mg) containing approximately 500-nCurie (nCi) of total radioactivity [14C]-ixazomib, solution, orally on Day 1 and ixazomib 4 mg, capsule, orally on Days 14 and 21 in Part A. Participants who had completed their Day 35 assessments in Part A were eligible to continue in Part B. Ixazomib 4 mg, capsule, orally, once weekly, on Days 1, 8 and 15 in 28-day cycles until disease progression or unacceptable toxicity in Part B.
Period: Overall Study
Arm/Group | Ixazomib
Started | 7
Completed | 5
Not Completed | 2
Not completed — Progressive disease | 2

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of ixazomib.
Arm/Group | Ixazomib
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (9.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1
  White | 5
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 164.4 (8.64)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 82.16 (16.772)

OUTCOME MEASURES:

1. Primary Outcome: Part A: Cmax: Maximum Observed Plasma Concentration for Ixazomib
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of ixazomib, obtained directly from the plasma concentration-time curve.
Time Frame: Day 1 of Part A pre-dose and at multiple timepoints (up to Day 14) post-dose
Population: Pharmacokinetic(PK)-evaluable population included all participants who received protocol-specified single[14C]-ixazomib dose(Part A), did not receive any excluded concomitant medications till completion(Part A), had sufficient concentration-time and total radioactivity(TRA)-time data to permit reliable estimation of PK parameters and mass balance.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Ixazomib
Number analyzed (Participants) | 5
nanogram per milliliter (ng/mL) | 89.06 (67.834)

2. Primary Outcome: Part A: Tmax: Time to Reach the Maximum Observed Plasma Concentration (Cmax) for Ixazomib
Description: Time to reach the maximum observed plasma concentration (Cmax), equal to time (hours) to Cmax of ixazomib after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Day 1 of Part A pre-dose and at multiple timepoints (up to Day 14) post-dose
Population: The PK-evaluable population included all participants who received the protocol-specified single [14C]-ixazomib dose in Part A, did not receive any excluded concomitant medications through the completion of Part A, and had sufficient concentration-time and TRA-time data to permit reliable estimation of PK parameters and mass balance.
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Ixazomib
Number analyzed (Participants) | 5
hour (hr) | 0.5000 (0.044721) [0.500 to 0.600]

3. Primary Outcome: Part A: AUC(0-312): Area Under the Plasma Concentration-time Curve From Time 0 to 312 Hrs Post-dose for Ixazomib
Description: AUC(0-312) is a measure of the area under the plasma concentration time-curve from time zero to 312 hrs post-dose for ixazomib.
Time Frame: Day 1 of Part A pre-dose and at multiple timepoints (up to 312 hrs) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Ixazomib
Number analyzed (Participants) | 5
nanogram*hour per milliliter (ng*hr/mL) | 1181 (600.53)

4. Primary Outcome: Part A: Cmax: Maximum Observed Plasma Concentration of TRA
Description: Maximum observed plasma concentration (Cmax) of TRA is the peak plasma concentration of TRA, obtained directly from the plasma TRA concentration-time curve.
Time Frame: Day 1 of Part A pre-dose and at multiple timepoints (up to Day 35) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: nanogram-equivalent per milliliter
Arm/Group | Ixazomib
Number analyzed (Participants) | 5
nanogram-equivalent per milliliter | 78.80 (48.814)

5. Primary Outcome: Part A: Tmax: Time to Reach the Cmax for TRA
Description: Time to reach the maximum observed plasma concentration (Cmax) for TRA, equal to time (hours) to Cmax for TRA after administration, obtained directly from the plasma TRA concentration-time curve.
Time Frame: Day 1 of Part A pre-dose and at multiple timepoints (up to Day 35) post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Ixazomib
Number analyzed (Participants) | 5
hr | 0.5000 (1.5547) [0.500 to 4.00]

6. Primary Outcome: Part A: AUC(0-816): Area Under the Plasma Concentration-time Curve From Time 0 to 816 Hrs Post-dose for TRA
Description: AUC(0-816) is a measure of the area under the plasma concentration time-curve from time zero to 816 hrs post-dose for TRA.
Time Frame: Day 1 of Part A pre-dose and at multiple timepoints (up to 816 hrs) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: nanogram-equivalent*hour per milliliter
Arm/Group | Ixazomib
Number analyzed (Participants) | 5
nanogram-equivalent*hour per milliliter | 2981 (1898.7)

7. Primary Outcome: Part A: Cmax: Maximum Observed Whole Blood Concentration of TRA
Description: Maximum observed whole blood concentration (Cmax) of a TRA is the peak whole blood concentration of TRA, obtained directly from the whole blood TRA concentration-time curve.
Time Frame: Day 1 of Part A pre-dose and at multiple timepoints (up to Day 35) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: nanogram-equivalent per milliliter
Arm/Group | Ixazomib
Number analyzed (Participants) | 5
nanogram-equivalent per milliliter | 181.6 (75.580)

8. Primary Outcome: Part A: Tmax: Time to Reach the Maximum Observed Whole Blood Concentration (Cmax) for TRA
Description: Time to reach the maximum observed whole blood concentration (Cmax) for TRA, equal to time (hours) to Cmax for TRA after administration, obtained directly from the whole blood TRA concentration-time curve.
Time Frame: Day 1 of Part A pre-dose and at multiple timepoints (up to Day 35) post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Ixazomib
Number analyzed (Participants) | 5
hr | 0.6000 (0.80436) [0.500 to 2.00]

9. Primary Outcome: Part A: AUC(0-816): Area Under the Whole Blood Concentration-time Curve From Time 0 to 816 Hrs Post-dose for TRA
Description: AUC(0-816) is a measure of the area under the whole blood concentration time-curve from time zero to 816 hrs post-dose for TRA.
Time Frame: Day 1 of Part A pre-dose and at multiple timepoints (up to 816 hrs) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: nanogram-equivalent* hour per milliliter
Arm/Group | Ixazomib
Number analyzed (Participants) | 5
nanogram-equivalent* hour per milliliter | 29200 (4712.2)

10. Primary Outcome: Part A: Cumulative Percentage of Ixazomib Dose Recovered in the Urine
Description: Percentage of the ixazomib dose excreted unchanged in the urine from 0 to 168 hrs post-dose.
Time Frame: Day 1 of Part A from 0 to pre-dose and at multiple timepoints (up to 168 hrs) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Ixazomib
Number analyzed (Participants) | 5
percentage of dose | 3.226 (2.1274)

11. Primary Outcome: Part A: Cumulative Percentage of the Total Radioactivity Dose Excreted in Feces
Description: Percentage of the TRA dose excreted in feces from Day 1 to Day 35 of Part A
Time Frame: Day 1 of Part A pre-dose and at multiple timepoints (up to Day 35) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Ixazomib
Number analyzed (Participants) | 5
percentage of dose | 21.80 (3.4147)

12. Primary Outcome: Part A: Cumulative Percentage of the Total Radioactivity Dose Excreted in Urine
Description: Percentage of the TRA dose excreted in urine from Day 1 to Day 35 of Part A.
Time Frame: Day 1 of Part A pre-dose and at multiple timepoints (up to Day 35) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Ixazomib
Number analyzed (Participants) | 5
percentage of dose | 62.06 (21.170)

13. Primary Outcome: Part A: Renal Clearance of Ixazomib
Description: Renal clearance is the volume of plasma from which ixazomib is completely removed by the kidney in a given amount of time, calculated as the amount of ixazomib excreted in the urine divided by the area under the plasma ixazomib concentration-time curve.
Time Frame: Day 1 pre-dose and at multiple timepoints (up to Day 14) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: liter per hour (L/hr)
Arm/Group | Ixazomib
Number analyzed (Participants) | 5
liter per hour (L/hr) | 0.1191 (0.068763)

14. Secondary Outcome: Ixazomib and Metabolites as Percent of Total Radioactivity in Plasma
Description: The plasma samples were pooled for participants over 816 hrs post-dose, and data was analysed using the Hamilton method time-proportional pooling, and therefore the data is reported as "percent of total radioactivity in plasma" with measure type as "number" and measure dispersion as "Not applicable, NA".
Time Frame: Day 1 pre-dose and at multiple time points (up to 816 hrs) post-dose
Population: PK-evaluable population with acceptable excretion recovery included all participants who received protocol-specified single[14C]-ixazomib dose(Part A), did not receive any excluded concomitant medications till completion(Part A), and had sufficient concentration-time and TRA-time data to permit reliable estimation of PK parameters and mass balance.
Measure: Number; unit: percent of total radioactivity in plasma
Arm/Group | Ixazomib
Number analyzed (Participants) | 4
percent of total radioactivity in plasma
  P4, ixazomib | 54.2
  P2, ML00701258 | 7.91
  P3, ML00701201 | 18.9
  P6, ML00749506 | 10.6
  P7, ML00752034 | 3.20

15. Secondary Outcome: Ixazomib and Metabolites as Percent of Total Dose Administered in Urine
Description: The 35-day post-dose data is extrapolated from the average of four participant data from 0-168-hr pooled urine. The data is therefore reported as "percentage of dose" with measure type as "number" and measure dispersion as "NA".
Time Frame: Day 1 pre-dose and at multiple time points (up to Day 35) post-dose
Population: as for outcome 14
Measure: Number; unit: percentage of dose
Arm/Group | Ixazomib
Number analyzed (Participants) | 4
percentage of dose
  U9, ixazomib | 1.30
  U1 | 0.391
  U2 | 0.926
  U3 | 1.61
  U4 | 1.33
  U5, ML00701258 | 2.72
  U6, ML00701201 | 30.2
  U7 | 2.75
  U8 | 0.695
  U10, ML00751996 | 5.93
  U11, ML00749506 | 1.28
  U12, ML00752034 | 0.069
  U13 | 0.974

16. Secondary Outcome: Ixazomib and Metabolites as Percent of Total Dose Administered in Feces
Description: The 35-day post-dose data is extrapolated from the average of four participant data from 0-168-hr pooled feces. The data is therefore reported as "percentage of dose" with measure type as "number" and measure dispersion as "NA".
Time Frame: Day 1 pre-dose and at multiple time points (up to Day 35) post-dose
Population: as for outcome 14
Measure: Number; unit: percentage of dose
Arm/Group | Ixazomib
Number analyzed (Participants) | 4
percentage of dose
  FH6, ixazomib | 13.8
  FH1 | 0.900
  FH2 | 0.111
  FH3, ML00701258 | 0.620
  FH4, ML00701201 | 0.901
  FH5 | 1.14
  FH7, ML00752034 | 1.58
  FH8 | 0.502
  FH9 | 0.112

17. Secondary Outcome: Number of Participants Reporting One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Baseline up to Cycle 5 Day 45
Population: The safety population included all participants who received at least 1 dose of ixazomib.
Measure: Number; unit: participants
Arm/Group | Ixazomib
Number analyzed (Participants) | 7
participants
  TEAEs | 7
  SAEs | 1

18. Secondary Outcome: Number of Participants With TEAEs Related to Investigations System Organ Class for Laboratory Values
Time Frame: Baseline up to Cycle 5 Day 45
Population: The safety population included all participants who received at least 1 dose of ixazomib.
Measure: Number; unit: participants
Arm/Group | Ixazomib
Number analyzed (Participants) | 7
participants
  Blood bilirubin increased | 1 (9.90)
  Platelet count decreased | 1 (25.53)
  Lymphocyte count decreased | 1 (117.64)

19. Secondary Outcome: Number of Participants With TEAEs Related to Vital Signs
Description: Vital signs included oral body temperature, heart rate, and blood pressure.
Time Frame: Baseline up to Cycle 5 Day 25
Population: The safety population included all participants who received at least 1 dose of ixazomib.
Measure: Number; unit: participants
Arm/Group | Ixazomib
Number analyzed (Participants) | 7
participants | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days after the last dose of study drug (Cycle 5 Day 45).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Ixazomib
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib (N=7)
Influenza (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib (N=7)
Diarrhoea (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Blood bilirubin increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Catheter site erythema (General disorders) | 1
Fatigue (General disorders) | 1
Gait disturbance (General disorders) | 1
Influenza like illness (General disorders) | 1
Malaise (General disorders) | 1
Medical device complication (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Drug hypersensitivity (Immune system disorders) | 1
Bladder spasm (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.